CLINICAL TRIAL: NCT05645016
Title: Church-Tailored Opioid Overdose Education and Naloxone Distribution to Target Overdose and Stigma Among African-American Communities
Brief Title: Tailoring Overdose Education for Black Churches
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The U.S. Department of Health and Human Services Office of Human Research Protections issued an FWA restriction on NYSPI research that included a pause of human subjects research as of June 23, 2023.
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Jermaine D. Jones, Associate Professor of Clinical Neurobiology, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 8208
Record Dates: First submitted 2022-11-30; First posted 2022-12-09 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Opioid Overdose
MeSH Terms: conditions — Opiate Overdose

STUDY DESIGN:
Intervention Model Description: The design is a two-arm cluster randomized trial with randomization at the level of the church (4 Churches), and analyses at the level of the individual participants (i.e., church members).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted Comprehensive Overdose Education and Skills Training (COEST) (Experimental)
  Interventions: Behavioral: COEST

INTERVENTIONS:
Behavioral: COEST — Adapted version of our COEST training, targeting Black church members.

SUMMARY:
Church-based interventions are culturally acceptable, reduce access barriers, and can be brought to scale in under-resourced communities. For Overdose Education and Naloxone Distribution (OEND) to be efficacious in Black churches, tailoring may be needed. For this audience, standard OEND curricula may need to be adapted to their level of knowledge of substance use disorders (SUDs), and limited general mental health literacy, and specifically address stigma related to SUDs and medications for opioid use disorder (MOUD). Finally, a tailored implementation strategy may need to address contextual variations (e.g., denomination and membership size) across churches. The proposed pilot study aims to identify the socio-cultural modifications that will be needed to adapt our previously developed training (i.e., COEST) to target Black communities of faith. In a pilot randomized controlled trial (RTC) of adapted COEST in a stepped-wedge design.

ELIGIBILITY:
Inclusion Criteria:

1. Identify as one of the following group members of the Black church: Clergy; Individual with OUD and/or stimulant use disorder; Family member or friend of an individual with OUD; Formerly incarcerated.
2. Age 18 and older.

Exclusion Criteria:

1. Unable to provide informed consent.
2. Less than 18 years old.
3. Does not identify as belonging to one of the four stakeholder groups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in Frequency of Naloxone Utilization/Overdose Intervention | Baseline and 6 Months after COEST training
  All study participants will receive an overdose response kit containing two doses of intranasal naloxone. Participants are asked to notify study staff immediately if they utilize naloxone in an attempt to reverse an opioid overdose.

SECONDARY OUTCOMES:
Opioid Overdose Knowledge Scale (OOKS) | Baseline and 6 Months after COEST training
  The OOKS measures knowledge about risk factors for having an opioid overdose, signs of an opioid overdose, actions to be taken in an overdose situation, naloxone effects and administration, adverse effects and aftercare procedures. The scale also identifies misinformation. The OOKS is a 14-item scale (Score Range: 0-45).
Brief Opioid Stigma Scale (BOOS) | Baseline and 6 Months after COEST training
  The BOSS was developed to assess stereotype awareness ("aware"), stereotype agreement ("agree"), and self-esteem decrement ("harm") surrounding opioid dependence. The BOSS is a 12-item scale (Score Range: 12-60)

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No